CLINICAL TRIAL: NCT05193630
Title: A Randomised, Open Label, Controlled Intervention Study to Investigate the Effects Oral Nutritional Supplement in Malaysian Children With Faltering Growth
Brief Title: Intervention Study to Investigate the Effects of ONS Use Among Malaysian Children With Faltering Growth
Acronym: MONS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Danone Specialized Nutrition (M) Sdn Bhd (Industry)
Collaborators: Universiti Putra Malaysia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FS21-MONS01
Record Dates: First submitted 2022-01-03; First posted 2022-01-18 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Faltering Growth
MeSH Terms: conditions — Failure to Thrive | interventions — Nutritional Support; Pharmaceutical Preparations

STUDY DESIGN:
Intervention Model Description: A randomised, open label, controlled intervention study
Who Masked: Outcomes Assessor
Masking Description: The anthropometric outcomes will be blinded to assessors and analyst until at least the primary outcomes have been analysed to reduce bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): The subjects in the treatment arm will be given Milnutri Sure TM product with dietary counselling
  Interventions: Dietary Supplement: Milnutri Sure™
- Control (Active Comparator): The subjects in the control arm, no Milnutri Sure TM product will be given, nevertheless, dietary counselling will be provided by the investigator.
  Interventions: Dietary Supplement: Milnutri Sure™

INTERVENTIONS:
Dietary Supplement: Milnutri Sure™ — Milnutri Sure™, a commercially available oral nutritional support (ONS) product in powder format, for children of 1 y of age and above (1.0 kcal /ml).
  For children between 1 and 3 years of age, the recommendation is to use 2 servings per day, and for children from 4 to 6 years of age, the recommendation is to give 3 servings per day. One serving contains of 45 grams of product and 180 ml water.
  Other Names: oral nutritional support (ONS) product in powder format

SUMMARY:
A randomised, open label, controlled intervention study to test the effect of the test product with dietary counselling versus dietary counselling alone on Weight-for-Age z-score change in children from ≥ 1 to ≤ 6 years of age with faltering growth for duration of 12 weeks.

DETAILED DESCRIPTION:
Parent(s) of potentially eligible subjects will be informed about the study and what is expected in case of participation to the study. Information on the study is incorporated in the Respondent's Information Sheet (RIS). The parent(s) will be given sufficient time to read and understand the Information Sheet and to ask questions. Parent(s) of eligible subjects will be approached at the main study clinic or they may be referred from one of the 'satellite clinics'. In case of referral, they will be pre-screened at the satellite clinic and if considered potentially eligible for the MONS study, they will be referred to the main study clinic for full screening.

If subjects fulfil all inclusion and exclusion criteria, and if the parent(s) is (are) willing that his/her/their child will participate, he/she/they will be asked to sign the Informed Consent Form (ICF). Baseline evaluation (including history and anthropometric measurement) will be completed prior to randomisation. A block randomisation will be performed to allocate subjects to treatment arm or control arm in 1:1 ratio.

At enrolment, the investigator assesses baseline characteristics, anthropometrics, appetite score, and the number of the child's sick days during the 4 weeks before enrolment. At the end of the visit, the investigator will provide two 3-days feeding diaries (one for baseline and one for Visit 2) and explain how and when these should be completed. The investigator will provide the Milnutri Sure™ product to the parent whose child is in the treatment arm, explain how to use the Milnutri Sure™ and how to apply other feeding advices for the coming 4 weeks until the next visit. For parent whose child is in the control arm, no Milnutri Sure TM product will be given, nevertheless, dietary counselling will be provided by the investigator.

Four, eight and twelve weeks after enrolment, subjects will have clinic visits (Visit 2, 3 and 4) and the anthropometrics, adverse events, appetite score, compliance, and the number of the children's sick days since last visit will be assessed. At the end of the visit the investigator will provide the product to the parents whose children are in the treatment arm, explains how to use it and how to apply other feeding advices for the coming 4 weeks until the next visit. For parents whose children are in the control arm, though no Milnutri Sure TM product will be given, dietary counselling will be provided by the investigator. At week eight (Visit 3), the investigator will also provide a 3-days feeding diary to the parents to be completed just before the twelve-week 12 visit (Visit 4).

In addition to this, at Visit 4 (the End of Study visit after 12 weeks in the study) the investigator will fill out the end of study visit requirements and stops providing study product. The investigator may request for a follow-up visit to monitor and provide medical and dietary counselling to the subject. If necessary, the investigator may prescribe Milnutri Sure ™ or any other growing up milk or nutritional counselling as part of normal practice.

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥1 and ≤ 6 years of age.
2. Weight at baseline between ≥ -3 and < -1 SD WHO-score (mild to moderate undernutrition).
3. Informed consent provided.

Exclusion Criteria:

1. Underlying medical illness affecting growth, according to the clinician's opinion
2. Known lactose intolerance / cow's milk allergy
3. Use of (other) ONS 1+ (1 kcal/mL) at enrolment and/or during the three months before enrolment
4. Other family member is already participating in this MONS study.
5. Insufficient ability to understand or communicate in English and/or Bahasa Malaysia
6. Participating in any other clinical study

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 172 (Estimated)
Dates: Start 2022-07-07 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
Weight for Age (WAZ) score of the subject | 12 weeks
  derived from weight and age

SECONDARY OUTCOMES:
Weight for Height (WHZ) score, weight and height of the subject | 12 weeks
  derived from height and weight
(Serious) Adverse Events of the IP and possible relatedness to study | 12 weeks
  Number, type and severity of (Serious) Adverse Events and possible relatedness to study product
Percentage of compliance | 12 weeks
  Percentage of compliance via missed servings compared to expected servings on product intake
Appetite score | 12 weeks
  Appetite score according to a visual analogue scale (0-10)
Nutritional intake | 12 weeks
  Total energy intake and nutrient intake from solid food

OTHER OUTCOMES:
Number of sick days | 12 weeks
  Number of sick days assessed via the investigator, who, at each clinic visit, asks the parents for the number of sick days during the past 4 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Zurina Zainudin, Principal Investigator — Universiti Putra Malaysia
Locations (1):
- Hospital Pengajar Universiti Putra Malaysia, Serdang, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No